CLINICAL TRIAL: NCT06076083
Title: Multicentar, Prospective Human Derived Materail Research for Two Group Cohort (Ankylosing Spondylitis Patient and Patient Family)
Brief Title: Multi-omics Database for Integrative Microbiome Analysis in a Cohort of Korean Patients With Ankylosing Spondylitis
Status: Recruiting | Type: Observational
Sponsor: Tae-Hwan Kim (Other)
Collaborators: Kyunghee University Medical Center (Other)
Responsible Party: Sponsor-Investigator, Tae-Hwan Kim, Professor, Hanyang University Seoul Hospital
Organization: Hanyang University Seoul Hospital (Other)
Other Study IDs: HI23C0661-MB-AS
Record Dates: First submitted 2023-09-20; First posted 2023-10-10 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-10

CONDITIONS: Ankylosing Spondylitis
Keywords: Microbiome; ankylosing spondylitis; multi-omics data
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — blood, saliva, feces, and intestinal mucosal tissue (patients who are scheduled for sigmoid colonoscopy or colonoscopy for routine examination) will be collected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ankylosing spondylitis patients: Ankylosing spondylitis Cohort consists of individuals aged 19 to 60 who, at the time of providing consent, have received a diagnosis of ankylosing spondylitis in accordance with the Modified New York criteria and meet the 2010 diagnosis of spondyloarthritis. These individuals have voluntarily chosen to participate in the study, having fully comprehended its details, and have agreed to adhere to the required precautions.
- ankylosing spondylitis patients their families: Those who are between the ages of 19 and 65 A primary immediate family member (parent/brother/sister) who is related to the patient and has never developed ankylosing spondylitis, and who lives with the patient 3) Those who, after listening to the explanation of this study and fully understanding it, voluntarily decided to participate and agreed to comply with the precautions

SUMMARY:
Multicenter Human Derivatives Prospective Cohort Study: Clinical information will be collected from patients with ankylosing spondylitis and their families who have provided research consent. And clinical samples including blood, saliva, feces, and mucosal biopsy tissue (from patients scheduled for sigmoid colonoscopy or routine colonoscopy examinations) will be collected. Multi-omics data production and laboratory analysis will be conducted using the collected samples, followed by integrated bioinformatic analysis using the produced data."

DETAILED DESCRIPTION:
Enrollment of ankylosing spondylitis patients and family controls who meet the exclusion criteria 2) Collection of standard clinical information items 3) Collect biological samples according to standardized protocols 4) Produce microbiome and multi-omics data from biosamples 5) Conduct clinical research using clinical information items and microbiome and multi-omics data

ELIGIBILITY:
Inclusion Criteria:

* Ankylosing spondylitis
* Age between 19 and 60 at the time of consent
* Diagnosis of ankylosing spondylitis based on the Modified New York criteria and the 2010 diagnosis of spondyloarthritis
* Willingness to participate voluntarily after comprehensively understanding the study and agreeing to adhere to the specified precautions

Family members of patients with ankylosing spondylitis

* Age between 19 and 65
* Must be a primary immediate family member (parent, brother, or sister) of the patient, who is related to the patient and has never been diagnosed with ankylosing spondylitis, and currently resides with the patient
* Willingness to participate voluntarily after attentively listening to the study's explanation, fully comprehending its details, and agreeing to adhere to the specified precautions

Exclusion Criteria for Ankylosing Spondylitis Patients:

1. Individuals who have taken antibiotics (oral/injected) within the last 3 months.
2. Individuals who have consumed lactic acid bacteria (health functional food) within the last 3 months.

Exclusion Criteria for Family Members of Ankylosing Spondylitis Patients:

Within a pre-planned period from the date of microbiome collection:

1. Individuals with a history of medication use listed in "drug use".
2. Individuals who have received a vaccine within the last 1 month (4 weeks) from the date of microbiome collection.
3. Individuals who have used topical antibiotics or topical steroids on the face, scalp, neck, arms, forearms, and hands within 24 hours of the date of microbiome collection.
4. Individuals who have used vaginal/vulvar medications, including antifungal drugs, within 24 hours from the date of microbiome collection.
5. Patients with acute illness (e.g., moderate or severe disease with or without fever, but sampling can be postponed until the subject recovers).
6. Patients with chronic and clinically significant medical conditions affecting the liver, digestive system, circulatory system, kidney, nervous system, respiratory system, endocrine system, immune system, blood system, malignant tumors, psychiatric history, or history of substance abuse.
7. Individuals who have made drastic changes to their diet for the purpose of rapid weight gain and loss within 4 weeks from the date of microbiome collection.
8. Individuals with gastrointestinal disorders that may affect microbiome analysis and are currently not medically controlled, or who are being treated for symptoms corresponding to the following diseases: Inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis), Irritable bowel syndrome (requiring medication), ulcers, acute or chronic pancreatitis, etc.
9. Individuals who need to use diapers for urinary incontinence.
10. Individuals who are suspected, based on medical opinion, to have conditions that may affect the collection of samples at the time of microbiome sample collection.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Depending on the contents of the Ministry of Health and Welfare's hospital-based human microbiome research and development project, the analysis method may change in the future.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Collect clinical information data for ankylosing spondylitis patients and their families | Visit 1 (0week)
  "Clinical information data will be collected from both ankylosing spondylitis patients and their families. Biosamples collected from these individuals will be used to establish a multi-omics analysis platform, including the examination of the intestinal microbiome. With this platform, comparative clinical studies will be conducted to uncover the disease's pathophysiology and identify potential biomarkers."

SECONDARY OUTCOMES:
Multi-omics data for ankylosing spondylitis patients and their families with consent. | Follow up Visit (24week)
  Diversity analysis: Alpha and beta diversity analyses are conducted to determine differences in the composition of gut microbiota between healthy individuals and patients.
  Important feature selection: Differential abundance analysis (e.g., using methods like LEfSe or ANCOM) or machine learning (e.g., random forest, support vector machine) is employed to identify microbiota.
  Functional profile prediction: In cases where metagenomic analysis is not feasible, the PICRUSt2 program is utilized to predict and analyze functional profiles based on the phylogeny of the microbiota present in healthy individuals and patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Hwan Kim, MD,PhD, Principal Investigator — Hanyang University Hospital for Rheumatic Diseases
Locations (2):
- South Korea (2):
  - Kyung Hee University Medical Center, Seoul, Kyungheedae-ro 23
  - Hanyang University Hospital for Rheumatic Diseases, Seoul, Wangsimni-ro222-1

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim HS, Kim BH, Nam B, Oh SJ, Park SK, Lee SW, Lee JY, Jo S, Lee YA, Lee JY, Park DI, Kim TH, Lee CK. Oral-gut microbiome axis in a Korean cohort with inflammatory bowel disease and ankylosing spondylitis (INTEGRATE): a prospective and observational study protocol. BMJ Open. 2025 Aug 10;15(8):e092075. doi: 10.1136/bmjopen-2024-092075. PMID 40784769